CLINICAL TRIAL: NCT06425237
Title: Evaluation of the Influence of Aromatherapy and Music Therapy on Stress During the Management of Cerebral Arteriography
Acronym: HERMES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/428/HP
Record Dates: First submitted 2024-04-09; First posted 2024-05-22 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Patients Scheduled for Cerebral Arteriography for Diagnostic or Therapeutic Purposes
MeSH Terms: interventions — Music Therapy; Aromatherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- standard care (No Intervention)
- standard care and music therapy (Experimental)
  Interventions: Other: music therapy
- standard care and aromatherapy (Experimental)
  Interventions: Other: aromatherapy
- standard care ansd music therapy and aromatherapy (Experimental)
  Interventions: Other: music therapy; Other: aromatherapy

INTERVENTIONS:
Other: music therapy — standard patient care in interventional radiology associated with a well-being atmosphere with the implementation of music therapy (soothing sound environment) in the preparation box and in the examination room.
  Arms: standard care and music therapy; standard care ansd music therapy and aromatherapy
Other: aromatherapy — standard patient care in interventional radiology associated with a well being atmosphere with the implementation of aromatherapy (essential oil of Ylang Ylang) in the preparation box and in the examination room.
  Arms: standard care and aromatherapy; standard care ansd music therapy and aromatherapy

SUMMARY:
Cerebral arteriography is a reference examination in medical imaging. This examination is performed to allow the diagnosis and therapeutic management of patients with vascular pathologies.

It is most often accompanied by a situation of stress, anxiety and apprehension related to the course of the examination or the announcement of the results.

These situations generate physiological reactions in patients, making the performance of cerebral arteriography more complex. In order to improve the quality of care for patients undergoing this invasive examination, it is proposed to use two non-medicinal techniques known for their soothing and relaxing properties: aromatherapy and music therapy alone or in combination. These two techniques will help to establish a common thread from the preparation of the patient before the examination to his return to the post-interventional surveillance room.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years old)
* Patient who is scheduled for a cerebral arteriography with local anaesthesia
* Patient who capable to read and understand the patient information and consent.
* Patient capable to read and sign the consent form
* Patient with social insurance
* Woman of childbearing age with effective contraception (see WHO definition), postmenopausal woman (≥ 12 months of amenorrhea not induced by therapy)
* Negative urine pregnancy test

Exclusion Criteria:

* Patients who have had a previous cerebral arteriogram
* Patient with allergy to iodinated contrast medium
* Patient with severe renal insufficiency
* Patient requiring sedation and artificial ventilation
* Patient who is deaf and/or hard of hearing
* Patient with a known allergy to essential oils
* Patient with anosmia

  * Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection, under guardianship or curatorship,
  * Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2027-11-04 (Estimated); Study Completion 2027-11-04 (Estimated)

PRIMARY OUTCOMES:
influence of aromatherapy and music therapy on the patient's stress when undergoing cerebral arteriography. | day 1
  blood pressure

SECONDARY OUTCOMES:
stress | day 1
  scale :0 : no stress to 10 : a lot of stress
level of pain | day 1
  scale : 0 : no pain to 10 : unbearable pain
hospital anxiety and depression scale | day 1
  scale : 0 to 7: no anxiety no depressed and 7 to 10 : probably anxiety ans drepressed more than and 10 : symptomatology of anxiety and depressed
Cumulative X-ray dose (mGy/cm2) received by the patient | day 1

CONTACTS AND LOCATIONS:
Overall Officials: Magali DUVAL, radiology technician, Principal Investigator — CHU Rouen
Locations (1):
- CHU de ROUEN, Rouen, France